CLINICAL TRIAL: NCT03567460
Title: Children and Adolescents With Marfan Syndrome: 10,000 Healthy Steps and Beyond
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Midwestern University (Other)
Responsible Party: Principal Investigator, Seda Tierney, Assistant Professor in Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 37176
Record Dates: First submitted 2017-10-03; First posted 2018-06-25 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Marfan Syndrome
MeSH Terms: conditions — Marfan Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10,000 Steps/day for Pediatric Marfan Patients (Experimental): Participants will be given a Garmin VivoFit and asked to take at least 10,000 steps per day. A study coordinator will reach out at least once per week to check in on progress made and help make weekly goals.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Across studies in adolescents in general population, 60 minutes of recommended daily exercise level is achieved, on average, within a total volume of 10,000-11,700 steps. The investigators will assess baseline physical activity quantitatively by using an accelerometer worn on the wrist during waking hours over a 7-day period. Each participant will be given a Garmin device to place on their wrist that will track their steps. Then patients will be asked to complete 10,000 steps daily for 6 months (acclimation over a week), which will be encouraged by daily text messages or e-mail, and weekly phone calls by the intervention team in addition to a Garmin and Facebook peer group.

SUMMARY:
Marfan patients are at risk of sudden death due to weakening of the wall of the large blood vessel leading from the heart (aorta). The wall of the aorta weakens and dilates which can rupture, leading to death, and sometimes during intense exercise.

There is some evidence in Marfan patients that a stiffer aorta increases risk for rupture.

For some time, clinical care has focused on what type of exercise these patients should avoid due to risk for aortic dissection. Little clinical emphasis has been placed on encouraging patients to engage in routine and safe exercise such as walking. Informed by this evidence, the investigators propose to collaboratively investigate whether regular exercise improves aortic health in adolescent Marfan patients.

DETAILED DESCRIPTION:
Marfan syndrome is an inherited disorder of the connective tissue, which provides material and support for the skeleton, muscles, and blood vessels. Marfan patients are at risk of sudden death due to weakening of the wall of the large blood vessel leading from the heart (aorta). The wall of the aorta weakens and dilates which can rupture, leading to death, and sometimes during intense exercise.

Typically, the weakening process starts when elastin fibers in the aorta become fragmented. There is some evidence in Marfan patients that a stiffer aorta increases risk for rupture.

For some time, clinical care has focused on what type of exercise these patients should avoid due to risk for aortic dissection. Little clinical emphasis has been placed on encouraging patients to engage in routine and safe exercise such as walking. These young patients also frequently choose sedentary lifestyles, most likely due to limitations imposed by parents as well as adolescents' own perceptions of what is safe for them and their physical capabilities. Another complicating factor is that these patients often experience difficulty coping with their diagnosis. Informed by this evidence, the investigators propose to collaboratively investigate whether regular exercise improves aortic health and coping skills in adolescent Marfan patients.

ELIGIBILITY:
Inclusion Criteria:

1. 10-19 years of age,
2. MFS by revised Ghent criteria,
3. Cardiac clearance to exercise by the primary cardiologist.

Exclusion Criteria:

1. Ventricular dysfunction,
2. Prior history of aortic surgery.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
To determine if 6 months of regular physical activity improves aortic stiffness in MFS patients. exercise, a decrease in expressed biomarkers, and an increase in COPE scores of MFS patients. | 6 months of intervention
  The investigators' primary outcome measure is aortic stiffness measured by arterial tonometry (pulse wave velocity).

SECONDARY OUTCOMES:
To determine if 6 months of regular physical activity improves aortic stiffness and the biomarker profile in MFS patients. | 6 months of intervention
  The secondary outcomes include aortic stiffness at the aortic root at the level of the sinuses of Valsalva and ascending aorta.
To determine if 6 months of regular physical activity improves aortic stiffness and the biomarker profile in MFS patients. | 6 months of intervention
  Secondary outcomes will be expression levels of TGF-β, Ang-II, MMP-2 & -9, ROS levels.
To determine if 6 months of regular physical activity decreases aortic stiffness and rate of aortic root dilation in Marfan mice. | 6 months of intervention
  Secondary outcomes will be expression levels of TGF-β, MMP-2, MMP-9, and ROS.
To determine if 6 months of regular physical activity improves coping skills in Marfan patients. | 6 months of intervention
  The outcome measure is the COPE inventory score.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Tierney, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Children's Health, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selamet Tierney ES, Chung S, Stauffer KJ, Brabender J, Collins RT 2nd, Folk R, Li W, Murthy AK, Murphy DJ, Esfandiarei M. Can 10 000 Healthy Steps a Day Slow Aortic Root Dilation in Pediatric Patients With Marfan Syndrome? J Am Heart Assoc. 2022 Dec 6;11(23):e027598. doi: 10.1161/JAHA.122.027598. Epub 2022 Dec 1. PMID 36453629